CLINICAL TRIAL: NCT04263909
Title: The Impact of Sublingual Sufentanil on Postoperative Pain and Analgesic
Brief Title: The Impact of Sublingual Sufentanil on Postoperative Pain and Analgesic Requirements in Spine Surgery Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Linda S Aglio, Associate Professor,, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020P000726
Record Dates: First submitted 2020-02-03; First posted 2020-02-11 (Actual); Results first posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Spine Fusion; Pain, Postoperative; Opioid Use
Keywords: sufentanil SL; Postoperative Pain; Spine Surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Administration, Sublingual; Sufentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- sufentanil SL arm (Experimental): Each patient will receive 30mcg of sufentanil SL prior to extubation in the operating room, and then as needed in the recovery room, guided by pain scores.
  Interventions: Drug: Sublingual Tablet

INTERVENTIONS:
Drug: Sublingual Tablet — sufentanil SL 30mcg administered sublingually to patients undergoing spine surgery before extubation and during recovery
  Other Names: sufentanil SL

SUMMARY:
In this study the investigators plan to examine the perioperative use of sufentanil sublingual (SL) in the analgesic regimen for spine surgery, one of the most common surgeries performed in the US. Patients undergoing spinal fusion surgery often experience severe pain during the first three postoperative days. Currently, no data are available for this patient population which routinely experiences moderate to severe acute pain. The investigators will analyze whether sufentanil SL is associated with lower opioid consumption in the post anesthesia care unit and pain scores.

DETAILED DESCRIPTION:
Sufentanil, unlike morphine and hydromorphone, avoids the issue of active metabolites that can lead to prolonged, untoward effects, which can complicate postoperative care and affect patient discharge. One study found that sufentanil SL 30 mcg was well tolerated, with no unexpected adverse events, no clinically meaningful vital sign changes, and a safety profile that was as expected for this postoperative patient population. In addition, the use of sufentanil SL in the emergency department indicates that sufentanil SL was a potentially feasible option for managing moderate-to-severe acute pain in that setting. Another study of adult patients undergoing major surgery in five hospitals in the Netherlands who received the sufentanil SL for postoperative pain relief as part of multimodal pain management showed that sufentanil SL effectively managed postoperative pain in abdominal and orthopedic surgeries. Finally, a randomized, open-label non-inferiority study that enrolled patients scheduled for elective major open abdominal or orthopedic surgery assessed the proportion of patients who responded "good" or "excellent" at the 48-hour timepoint on the Patient Global Assessment of method of pain control. The results showed that 78.5% vs. 65.6% of patients achieved "success" for sufentanil SL vs. intravenous patient-controlled analgesia (morphine), respectively, demonstrating non-inferiority as well as statistical superiority for treatment effect. Patients using sufentanil SL reported more rapid onset of analgesia and patient and nurse ease of care and satisfaction scores were higher than intravenous patient-controlled analgesia (morphine). Adverse events were similar between the 2 groups, and sufentanil SL had fewer patients experiencing oxygen desaturations below 95% compared to intravenous patient-controlled analgesia (morphine). Future studies are needed to determine patient populations that benefit most from the sufentanil SL, assess the added values versus intravenous patient-controlled analgesia, and determine the pharmacoeconomics of the system.

Purpose:

In this study the investigators plan to examine the perioperative use sufentanil SL in the analgesic regimen for spine surgery, one of the most common surgeries performed in the United States. Patients undergoing spinal fusion surgery often experience severe pain during the first three postoperative days. Currently, no data are available for this patient population which routinely experiences moderate to severe acute pain. The investigators will analyze whether sufentanil SL is associated with lower opioid consumption, number of fentanyl boluses given, post-anesthesia care unit and hospital length of stay, side effects of opioid use (i.e., nausea, vomiting, constipation), and hospitalization costs (i.e., pharmacoeconomics).

Hypotheses:

1. The perioperative use of sufentanil SL 30 mcg in a prospective cohort of patients undergoing spine surgery will be associated with lower postoperative numeric rating scale pain scores (numerical rating score (NRS); primary outcome) than observed in two historical control groups that did not receive sufentanil SL: one group that received intraoperative remifentanil infusion and one that received intraoperative sufentanil infusion.
2. The perioperative use of sufentanil SL will be associated with lower opioid consumption, number of fentanyl boluses given, post-anesthesia care unit length of stay than observed in two historical control groups of patients receiving remifentanil or sufentanil infusions without perioperative sufentanil SL.

Methods:

The study design is a prospective cohort study with historical controls. There will be 1 prospectively recruited study arm (30 patients receiving the study drug sufentanil SL) and 2 historical control arms (one that received an intraoperative remifentanil infusion, 80 patients, and the other that received an intraoperative sufentanil infusion, 80 patients, both without sufentanil SL).

Inclusion criteria include patients undergoing spine surgery (1- 3 levels) who are opioid-naïve, 18-75 years old, considered American Society of Anesthesiologists (ASA) physical status 1-3 and also includes patients with impaired renal function.

Exclusion criteria include those with microdiscectomy, have chronic opiate use, significant respiratory depression, acute or severe bronchial asthma, chronic lung disease, known or suspected gastrointestinal obstruction including paralytic ileus, liver disease ((defined as alkaline phosphatase (ALP) > 56, aspartate aminotransferase (AST)> 100), known allergy or hypersensitivity to sufentanil or its components, baseline dementia, serotonin syndrome, adrenal insufficiency, severe hypotension, increased intracranial pressure, brain tumors, head injury, impaired consciousness, malignant hyperthermia, ASA physical status >3, age >75, and pregnant patients.

Outcomes:

Primary:

Pain scores in post-anesthesia care unit (PACU)

Secondary:

Length of stay: PACU Length of stay: inpatient Hospital stay Pain scores: inpatient Hospital stay Opioid consumption: PACU Opioid consumption: inpatient Hospital stay

As shown above, the above primary and secondary outcomes will also be collected in the prospective cohort to obtain estimates that can be used to power future randomized controlled trials.

Safety assessments will include adverse events and use of concomitant medications, periodic monitoring of vital signs (blood pressure, heart rate, and respiratory rate), and continuous monitoring of oxygen saturation in the post-anesthesia care unit.

Intraoperative Management:

The prospective study arm will receive general endotracheal anesthesia consisting of total intravenous anesthesia maintained with continued infusions of propofol (80-200 mcg/kg/min) and sufentanil (0.2-0.3mcg/kg/hr). Anesthesia induction will be achieved with propofol (1.5-2.5mg/kg), succinylcholine (1mg/kg), and sufentanil (10-20 mcg). The study group will receive sufentanil SL 30 mcg at surgery end, but prior to emergence from anesthesia, and after the patient is turned supine. Antiemetic prophylaxis will be administered (ondansetron).

Postoperative Management:

Note that sufentanil SL will be ordered as q1hr prn, meaning that repeat doses must be administered at least 1 hr apart.

In the post-anesthesia care unit, patients will be ordered to receive sufentanil SL 30 mcg prn 1 hr for breakthrough pain (for numerical rating scale, NRS > 3) as the 1st line analgesic, with hydromorphone as the rescue analgesic if the patient is still experiencing pain (NRS >3). The following opioid administration schema will be used for pain management in the post-anesthesia care unit:

* 1st line: sufentanil SL 30mcg (NRS >3). 2nd line: hydromorphone 0.2-0.6 mg (NRS >3)
* If upon arrival to the PACU the patient is still experiencing pain with NRS >3 but cannot yet receive a repeat dose of sufentanil SL (because of having received 1st dose in the operating room less than 1 hour ago), then the patient can receive hydromorphone 0.2-0.6 mg prn until eligible to receive sufentanil SL.
* If at any time the patient's NRS >3 after 20 min following an administration of either sufentanil SL or fentanyl, the patient can receive a repeat dose of fentanyl until again eligible to receive sufentanil SL.

Once the patient is transferred to the floor, both groups will receive the standard of care postoperative pain management orders (ie oral and intravenous prn analgesia for NRS > 3).

Sample Size/Statistical analysis:

Assuming a within-group standard deviation in post-anesthesia care unit NRS pain score of 2.5 points, enrollment of 30 patients in the prospective group and inclusion of at least 80 patients in each retrospective control group will provide at least 80% power at a two sided alpha level of 0.025 (0.05/2 pair-wise comparisons) to detect a minimal clinically important difference of 2 points between the prospective group and each of the retrospective groups using linear regression.

All outcomes will be compared between the prospective group and each of the retrospective groups using linear regression weighted by inverse probability of treatment weights. Probability of treatment (i.e., propensity scores) will be calculated using logistic regression with the following covariates: age, sex, body mass index, American Society of Anesthesiologists class, surgical invasiveness tier, reoperation, history of anxiety, anxiolytic use, history of depression, and antidepressant use.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing spine surgery (> 1 levels)
* Opioid-naïve
* ≥18 years old
* American Society of Anesthesiologists class 1-4
* Planned inpatient stay

Exclusion Criteria:

* Microdiscectomy or single level surgery
* Chronic opiate use
* Liver disease
* Allergy/hypersensitivity to sufentanil
* Patients with baseline dementia
* Plan outpatient surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2023-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard D. Urman, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bernstein MH, Beaudoin FL, Magill M. Response to FDA Commissioner's statement on Dsuvia approval. Addiction. 2019 Apr;114(4):757-758. doi: 10.1111/add.14539. Epub 2019 Jan 20. No abstract available. PMID 30589478
- [Background] Sufentanil. 2025 Dec 15. Drugs and Lactation Database (LactMed(R)) [Internet]. Bethesda (MD): National Institute of Child Health and Human Development; 2006-. Available from http://www.ncbi.nlm.nih.gov/books/NBK501254/ PMID 30000313
- [Background] van de Donk T, Ward S, Langford R, Dahan A. Pharmacokinetics and pharmacodynamics of sublingual sufentanil for postoperative pain management. Anaesthesia. 2018 Feb;73(2):231-237. doi: 10.1111/anae.14132. Epub 2017 Dec 8. PMID 29219169
- [Background] Babazade R, Turan A. Sufentanil sublingual tablet system for the management of postoperative pain. Expert Opin Pharmacother. 2016 Dec;17(17):2351-2357. doi: 10.1080/14656566.2016.1254190. PMID 27796147
- [Background] Deeks ED. Sufentanil 30 microg Sublingual Tablet: A Review in Acute Pain. Clin Drug Investig. 2019 Apr;39(4):411-418. doi: 10.1007/s40261-019-00772-x. PMID 30887417

RESULTS

PARTICIPANT FLOW:
Groups:
- Sufentanil SL Arm: Each patient received 30mcg of sufentanil SL prior to extubation in the operating room, and then as needed in the recovery room, guided by pain scores.
  Sublingual Tablet: sufentanil SL 30mcg administered sublingually to patients undergoing spine surgery before extubation and during recovery
- IV Remifentanil Historical Arm: Each patient received intraoperative remifentanil and hydromorphone for postoperative pain
- IV Sufentanil Historical Arm: Each patient received intraoperative sufentanil and hydromorphone for postoperative pain
Period: Overall Study
Arm/Group | Sufentanil SL Arm | IV Remifentanil Historical Arm | IV Sufentanil Historical Arm
Started | 39 | 80 | 80
Completed | 30 | 80 | 80
Not Completed | 9 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Adverse Event | 3 | 0 | 0
Not completed — Protocol Violation | 5 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sufentanil SL Arm | IV Remifentanil Historical Arm | IV Sufentanil Historical Arm | Total
Number analyzed (Participants) | 30 | 80 | 80 | 190
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (14.2) | 57.0 (11.3) | 58.8 (12.4) | 58.0 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 49 | 43 | 107
  Male | 15 | 31 | 37 | 83
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4 | 8
  Not Hispanic or Latino | 28 | 76 | 75 | 179
  Unknown or Not Reported | 1 | 1 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 5 | 5 | 10
  White | 27 | 72 | 72 | 171
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 3 | 9
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.9 (6.9) | 29.6 (5.1) | 29.3 (5.9) | 29.5 (5.7)
ASA Class [Count of Participants; unit: Participants] — The American Society of Anesthesiologists physical status classification system provides perioperative clinicians with a standardized method to evaluate a patient's medical comorbidities & help predict perioperative risk. It consists of 6 ordinal scoring categories (and one additional designation for emergencies) to succinctly communicate a general assessment of underlying physiologic status, ranging from completely healthy (ASA Class I) to brain-dead awaiting organ procurement for donation (ASA Class VI).
  Participants
    Class 1 (Normal healthy patient, no systemic disease) | 1 | 0 | 2 | 3
    Class 2 (mild systemic disease with no functional limitations | 7 | 32 | 36 | 75
    Class 3 (severe systemic disease that may limit activity or function but is not a threat to life) | 22 | 48 | 42 | 112
Surgical Invasiveness Tier [Count of Participants; unit: Participants] — The surgical invasiveness tier system categorizes spinal surgeries as follows with tier 1: microdiscectomy, tier 2: lumbar laminectomy, anterior cervical procedures, or minimally invasive spinal fusions, tier 3: standard or complex lumbar fusion, emergency surgery following trauma, or posterior cervical fusion procedures, and tier 4: surgeries to ameliorate tumor, infection, or deformity, or combined anterior and posterior cervical procedures.
  Participants
    tier 1: microdiscectomy | 2 | 0 | 5 | 7
    tier 2: lumbar laminectomy, anterior cervical procedures, or minimally invasive spinal fusions | 18 | 36 | 42 | 96
    tier 3: standard/complex lumbar fusion, emergency surgery following trauma posterior cervical fusion | 8 | 40 | 30 | 78
    tier 4: surgeries to remove tumor, infection/deformity, or combined anterior & posterior cervical . | 2 | 4 | 3 | 9
History of Anxiety [Count of Participants; unit: Participants] | 9 | 20 | 19 | 48
Anxiolytic Use [Count of Participants; unit: Participants] | 2 | 13 | 11 | 26
History of Depression [Count of Participants; unit: Participants] | 7 | 11 | 15 | 33
Antidepressant Use [Count of Participants; unit: Participants] | 5 | 18 | 15 | 38
Surgery duration (minutes) [Median (Inter-Quartile Range); unit: minutes] | 182.5 [156.3 to 227] | 224.0 [176.8 to 292.0] | 249.0 [200.5 to 328.0] | 229.0 [176.2 to 307.8]
Intraoperative IV acetaminophen [Count of Participants; unit: Participants] | 20 | 43 | 28 | 91
Average PACU pain score [Mean (Standard Deviation); unit: units on a scale] — NSR or numeric pain rating scale is a pain assessment tool where patients rate their pain level on a scale of 0 to 10, with 0 representing no pain and 10 representing worst possible pain. Interpretation of the score, 0=no pain, 1-3 = mild pain, 4-6 = moderate pain and 7-10 = severe pain.
  units on a scale | 3.2 (2.4) | 5.7 (2.2) | 5.0 (2.4) | 5.0 (2.4)

OUTCOME MEASURES:

1. Primary Outcome: Average Postoperative Pain Score - PACU/ Post-anesthesia Care Unit
Description: pain scores as reported by the patient using NRS (numerical rating scale) 0 (no pain)-10 (worst possible pain)
Time Frame: Up to 120 minutes after arrival to PACU
Measure: Mean (Standard Deviation); unit: Pain score NSR
Arm/Group | Sufentanil SL Arm | IV Remifentanil Historical Arm | IV Sufentanil Historical Arm
Number analyzed (Participants) | 30 | 80 | 80
Pain score NSR | 3.22 (2.42) | 5.66 (2.19) | 5.05 (2.38)

2. Secondary Outcome: Opioid Consumption - PACU
Description: total amount of opioids (in morphine milligram equivalents) used
Time Frame: up to 120 min after arrival to the post anesthesia care unit (PACU)
Measure: Mean (Standard Deviation); unit: morphine milligram equivalents
Arm/Group | Sufentanil SL Arm | IV Remifentanil Historical Arm | IV Sufentanil Historical Arm
Number analyzed (Participants) | 30 | 80 | 80
morphine milligram equivalents | 6.13 (10.79) | 29.02 (21.45) | 23.06 (21.61)

3. Secondary Outcome: Opioid Consumption - Inpatient Floor
Description: total amount of opioids (in morphine milligram equivalents) used
Time Frame: up to 48 hours, from arrival to inpatient floor until discharge home
Measure: Mean (Standard Deviation); unit: morphine milligram equivalents
Arm/Group | Sufentanil SL Arm | IV Remifentanil Historical Arm | IV Sufentanil Historical Arm
Number analyzed (Participants) | 30 | 80 | 80
morphine milligram equivalents | 41.59 (36.43) | 74.51 (44.17) | 74.99 (45.71)

4. Secondary Outcome: Postoperative Pain Scores - Inpatient Floor
Description: pain scores as reported by the patient using NRS (numerical rating scale) 0 (no pain)-10 (worst possible pain)
Time Frame: up to 48 hours, from arrival to inpatient floor until discharge home
Measure: Mean (Standard Deviation); unit: Pain score NSR
Arm/Group | Sufentanil SL Arm | IV Remifentanil Historical Arm | IV Sufentanil Historical Arm
Number analyzed (Participants) | 30 | 80 | 80
Pain score NSR | 3.96 (1.61) | 4.84 (1.55) | 4.54 (1.37)

5. Secondary Outcome: Length of Stay in the PACU
Description: the amount of time (in minutes) the patient stayed in the PACU until the patient was signed out as ready to be transferred to inpatient floor
Time Frame: up to 24 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sufentanil SL Arm | IV Remifentanil Historical Arm | IV Sufentanil Historical Arm
Number analyzed (Participants) | 30 | 80 | 80
minutes | 129.23 (77.15) | 127.53 (54.83) | 118.50 (52.59)

6. Secondary Outcome: Length of Stay on the Inpatient Floor
Description: the amount of time (in days) the patient stayed on the inpatient floor until the patient was discharged to home
Time Frame: up to 30 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Sufentanil SL Arm | IV Remifentanil Historical Arm | IV Sufentanil Historical Arm
Number analyzed (Participants) | 30 | 80 | 80
days | 1.11 (0.74) | 2.09 (1.78) | 2.19 (1.67)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored during the first two hours of the patient's post operative period of recovery.
Description: Nausea or vomiting within the first two hours of taking SST
Arm/Group | Sufentanil SL Arm | IV Remifentanil Historical Arm | IV Sufentanil Historical Arm
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/80 | 0/80
Serious Adverse Events (participants affected / at risk) | 3/39 | 0/80 | 0/80
Other Adverse Events (participants affected / at risk) | 0/39 | 0/80 | 0/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sufentanil SL Arm (N=39) | IV Remifentanil Historical Arm (N=80) | IV Sufentanil Historical Arm (N=80)
Other (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) — Patients sensitive to medication

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-28): https://cdn.clinicaltrials.gov/large-docs/09/NCT04263909/Prot_SAP_000.pdf